CLINICAL TRIAL: NCT06494046
Title: Defining Musical Toxicity and Its Effect on Patient Well-being
Status: Withdrawn | Type: Observational
Why Stopped: Resident working with study left institution
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR2333; NCI-2024-05423 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-012760 (Other: Mayo Clinic Institutional Review Board); ROR2333 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Esophageal Carcinoma; Head and Neck Carcinoma; Lung Carcinoma; Malignant Brain Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Esophageal Neoplasms; Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observational Musical Toxicity Group: Patients complete a questionnaire, participate in an interview and their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Observational No Musical Toxicity Group: Patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates the experience of musicians who are going through cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe specific musical difficulties that arise during and after cancer treatments: define "musical toxicity".

II. Discover any interventions or treatments which musicians found helpful while going through cancer treatment.

III. Investigate whether the priority of playing music changed through the course of cancer treatment and beyond, in relation to other priorities including cancer cure and length of life.

IV. Discover treatment and cancer related factors which are correlated with worse musical toxicity.

OUTLINE: This is an observational study. Patients are assigned to 1 of 2 groups.

MUSICAL TOXICITY GROUP: Patients complete a questionnaire, participate in an interview and have their medical records reviewed on study.

NO MUSICAL TOXICITY GROUP: Patients have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Adults ≥ 18 years or older

  * Active or accomplished musicians

    * Those performing in the community as part of a group or as a soloist
    * Those teaching lessons in an individual or group setting
    * Those for whom music teaching or performance is a primary source of income
    * Those who play music multiple times per week
  * Our ideal cohort will consist of an equal number of patients with the following malignancies above the diaphragm:

    * Brain
    * Head and Neck
    * Esophagus or Lung
    * Breast
  * Our ideal cohort will consist of an equal number of patients who engage in the following musical endeavors:

    * Stringed instruments
    * Wind instruments (including woodwind and brass instruments)
    * Keyboard instruments
    * Vocalists

Exclusion Criteria:

* * < 18 years

  * Did not regularly attempt to engage in musical endeavors during or after cancer treatment
  * Not willing or able to complete the questionnaire or engage in a one-hour interview (i.e. limited English proficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are active or accomplished musicians undergoing cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Describe specific musical difficulties that arise during and after cancer treatments - MTQ 10-item | Baseline
  Assessed using the Musical Toxicity Questionnaire (MTQ 10-item), a survey with yes/no and open-ended questions (e.g., What musical instrument do you play, or do you sing?). The survey is designed to capture the participant's thoughts and feelings on how cancer treatments (before and after) has affected enjoyment and ability to play, teach, or perform music. The questionnaire will take about 15-30 minutes to complete. Qualitative analysis software will be utilized to code responses and organize themes. Themes will be organized into related groups and interpreted to generate conclusions.

CONTACTS AND LOCATIONS:
Overall Officials: Dean A. Shumway, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials